CLINICAL TRIAL: NCT07394647
Title: Transcutaneous Auricular Vagus Nerve Stimulation for Preventing Emergence Agitation and Delirium After Pediatric Tonsillectomy and Adenoidectomy: A Randomized, Double-Blind, Interventional Study
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation for Prevention of Emergence Agitation and Delirium in Children Undergoing Tonsillectomy and Adenoidectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MR-33-25-067114
Record Dates: First submitted 2025-12-10; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-02

CONDITIONS: Emergence Agitation; Emergence Delirium
Keywords: Pediatric; Emergence Agitation; Emergence Delirium; taVNS; Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the active transcutaneous auricular vagus nerve stimulation (taVNS) group or the sham stimulation group. Both participants and study personnel involved in intervention delivery and outcome assessment are blinded to group allocation. The effects of taVNS on emergence agitation and emergence delirium after pediatric tonsillectomy and adenoidectomy will be compared between the two parallel groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active taVNS Group (Experimental): Participants in this group will receive active transcutaneous auricular vagus nerve stimulation (taVNS) during the perioperative period.
  Stimulation will be applied to the left cymba conchae using an ear-clip electrode connected to a portable taVNS device.
  Parameters: 25 Hz frequency, 300 µs pulse width, duty cycle 30 seconds ON / 30 seconds OFF.
  The stimulation starts before anesthesia induction and continues during surgery and recovery in the PACU.
  On postoperative days 1 and 2, stimulation will be administered twice daily for 30 minutes each session.
  Intensity is adjusted until a mild tingling sensation is perceived without pain.
  Interventions: Device: Active taVNS Group
- Sham Stimulation Group (Sham Comparator): Participants receive sham stimulation applied to the left auricular concha. The device is applied in the same manner as the active group, but stimulation is inactive after initial titration. Stimulation schedule and duration are identical to the active group to maintain blinding
  Interventions: Device: Sham stimulation group

INTERVENTIONS:
Device: Active taVNS Group — Active taVNS Group：The taVNS device delivers electrical stimulation via an ear-clip electrode placed on the left cymba conchae.Parameters: 25 Hz frequency, 300 µs pulse width, 30 s ON / 30 s OFF duty cycle.Applied from pre-induction through postoperative recovery, then twice daily for 30 min on POD 1-2.Intensity adjusted to induce mild tingling without discomfort.
  Arms: Active taVNS Group
Device: Sham stimulation group — The sham stimulation device is visually identical to the active taVNS unit. Electrodes are placed on the same auricular site, and procedures mimic active stimulation, but no electrical current is delivered.Used to maintain blinding and control for placebo effects.
  Arms: Sham Stimulation Group

SUMMARY:
Brief Summary This study is designed to find out whether transcutaneous auricular vagus nerve stimulation (taVNS) can safely reduce restlessness and confusion when children wake up from anesthesia after tonsillectomy and adenoidectomy. These problems, called emergence agitation and delirium, are common after surgery and can cause distress for both children and their families.TaVNS is a non-invasive treatment that delivers mild electrical stimulation to a specific area of the ear connected to the vagus nerve. It does not involve needles or medication, and children usually feel only a gentle tingling sensation.In this randomized, double-blind study, children will be assigned by chance to receive either taVNS or a sham (placebo) stimulation during surgery. Neither the children, their families, nor the medical team providing care will know which treatment each child receives.Researchers will observe and record how calmly children wake up from anesthesia, whether they show signs of delirium, and any side effects. The goal of this study is to test whether taVNS is an effective and safe way to improve recovery and comfort for children after surgery.

DETAILED DESCRIPTION:
Background and Rationale Emergence delirium (ED) in pediatric patients is a common postoperative complication linked to exposure to volatile anesthetics, particularly sevoflurane. The proposed mechanism involves dysregulation of the autonomic nervous system, characterized by reduced vagal tone and sympathetic hyperactivity. Transcutaneous auricular vagus nerve stimulation (taVNS) is a non-invasive neuromodulation technique designed to increase vagal activity by delivering low-intensity electrical currents to the auricular branch of the vagus nerve in the ear. Preclinical and clinical evidence suggests taVNS can exert anti-inflammatory, analgesic, and anxiolytic effects via central and peripheral pathways. This trial is designed to investigate whether perioperative taVNS can mitigate ED by modulating autonomic balance.

Intervention and Blinding Methodology The study employs a double-blind, sham-controlled design. Active and sham stimulation devices are physically identical. The active device delivers electrical stimulation with parameters set at a frequency of 25 Hz, a pulse width of 300 μs, and a cyclic mode of 30 seconds on followed by 30 seconds off. Stimulation intensity is individually titrated to a perceptible but non-painful tingling sensation. The sham device follows an identical placement and titration procedure but ceases output after the initial adjustment phase. This methodology ensures participants, caregivers, and outcome assessors are blinded to group assignment. Stimulation is initiated in the preoperative holding area, continues intraoperatively, and concludes upon discharge from the post-anesthesia care unit (PACU). Supplemental stimulation sessions are administered on postoperative days 1 and 2.

Study Procedures Overview Following enrollment and randomization, the stimulation device is applied to the left auricular concha. Standardized general anesthesia is administered per protocol, utilizing sevoflurane for maintenance with titration guided by bispectral index (BIS) monitoring. Intraoperative vital signs and anesthetic depth are recorded. Upon cessation of anesthetics, continuous behavioral observation begins in the PACU.

Technical and Mechanistic Considerations The selection of the left auricle for stimulation is based on anatomical studies indicating a lower density of cardiac vagal fibers compared to the right side. The chosen stimulation parameters (25 Hz, 300 μs) are derived from prior neurophysiology studies suggesting efficacy in activating afferent vagal pathways. The cyclic on/off pattern is intended to prevent nerve accommodation. The perioperative timing of stimulation is designed to preemptively modulate autonomic tone prior to the emergence phase, a period of high neurophysiological lability.

Data Collection and Management Primary and secondary outcome data are collected at predetermined time points by trained, blinded assessors. Data pertaining to device adherence (session timing, wear status) are recorded by nursing staff. All data are entered into a secure, electronic data capture system. Source data verification is performed per the monitoring plan.

Statistical Considerations The primary analysis will utilize the intention-to-treat principle. The primary endpoint, incidence of emergence delirium, will be compared between groups using a chi-square test. A secondary logistic regression analysis will adjust for predefined covariates (e.g., age, surgery duration) to evaluate the independent effect of the intervention. Analysis of continuous secondary endpoints will employ t-tests or non-parametric equivalents based on data distribution. A two-sided p-value <0.05 will define statistical significance.

Safety Monitoring Adverse events are monitored from device application through the follow-up period. Specific attention is given to local skin reactions at the electrode site and any potential device-related incidents. All adverse events are documented and reported according to the protocol and regulatory requirements.

Significance and Implications This investigation aims to provide high-level evidence on the efficacy of a non-pharmacologic, neuromodulatory approach to preventing pediatric emergence delirium. Positive results could establish taVNS as a viable strategy to enhance postoperative recovery and safety, with potential implications for broadening the application of bioelectronic medicine in perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 8 years.
* Patients receiving care at The First Affiliated Hospital of Zhejiang Chinese Medical University with a diagnosis of tonsil and/or adenoid hypertrophy, scheduled for tonsillectomy and/or adenoidectomy under sevoflurane inhalation general anesthesia.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Ability to understand the study procedures and assessment scales, and to communicate effectively with study personnel.

Exclusion Criteria:

* ASA physical status III-IV, or presence of hepatic or renal dysfunction, cardiovascular disease, or endocrine disorders.
* Neuromuscular disorders or dermatitis of the left auricle.
* Recent respiratory infection, developmental delay, or autism spectrum disorder.
* Receipt of specialized care, residence in social welfare institutions, or any other condition that may interfere with study participation.
* Current enrollment in another clinical trial.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of emergence delirium (ED) | Every 10 min during after the patient removed the endotracheal tube ，in the first 30 min in the Post-Anesthesia Care Unit (PACU).
  Measurement Tools: Diagnosis will be made using the Pediatric Anesthesia Emergence Delirium (PAED) Scale (score range: 0-20, higher scores indicate worse delirium) and the FLACC (Face, Legs, Activity, Cry, Consolability) Pain Scale (score range: 0-10, higher scores indicate worse pain).
  Diagnostic Criteria:
  1. ED is defined as a PAED score ≥ 10 and a FLACC score < 4.
  2. If both PAED score ≥ 10 and FLACC score ≥ 4, the child will first receive intravenous fentanyl 0.5 μg·kg-¹ for analgesia.
  3. Five minutes after analgesia, both scales will be reassessed. If the PAED score remains ≥ 10, the diagnosis of ED will be confirmed regardless of the FLACC score.

SECONDARY OUTCOMES:
The incidence of postoperative pain | Assessed at 0, 5, 10, 20, and 30 minutes after emergence from anesthesia.
  Defined as a FLACC score (Face, Legs, Activity, Cry, Consolability scale; score range 0-10, where higher scores indicate worse pain outcomes) of ≥ 4.
Quality of Recovery in Children (PedS-QoR Score) | Assessed at 24 and 48 hours after surgery.
  Postoperative recovery quality will be assessed using the Pediatric Quality of Recovery Scale (PedS-QoR, 20-item version).
  This validated questionnaire evaluates children's physical comfort, emotional state, psychological well-being, and independence after surgery and anesthesia.
  Proxy Report: For children aged 2-7 years, completed by parents or caregivers. Self-Report: For children aged 8-17 years, completed by the child. The total score ranging from 20 to 100, where higher scores indicate better recovery quality.
Recovery Time | Recovery parameters were assessed every 5 min in the first 30 min after anesthesia discontinuation and then every 10 min until discharge criteria were met or up to 120 min.
  The time interval from the discontinuation of sevoflurane to the moment when the child is awakened and able to respond to their name spoken in a normal tone of voice, including cases where response is delayed due to emergence delirium (ED).
Adverse Events | From initiation of the intervention through 3 days after surgery.
  All adverse events occurring during hospitalization will be recorded, including nausea, vomiting, pneumonia, and ta-VNS-related complications such as skin irritation, dizziness, or bradycardia.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang Chinese Medical University (Zhejiang Provincial Hospital of Traditional Chinese Medicine), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available beginning 6 months after publication of the primary results manuscript. Data will be shared with researchers who provide a methodologically sound proposal for use in non-commercial research. Proposals should be directed to the corresponding author. To gain access, requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Supporting information (study protocol and statistical analysis plan) will be available beginning 6 months after study completion and for up to 3 years following publication of the primary results.
Access Criteria: Access to the study protocol and statistical analysis plan will be granted to academic researchers affiliated with recognized institutions for non-commercial research purposes. Requests should be submitted to the principal investigator by email. Data sharing will require prior approval and signing of a data use agreement.

REFERENCES:
- [Background] Graydon C, Stricker PA, Kelleher S, Cravero J, Karim N, Muhly WT, Lee-Archer P. Development of the Pediatric Scale for Quality of Recovery (PedSQoR). Anesthesiology. 2025 Aug 1;143(2):275-286. doi: 10.1097/ALN.0000000000005503. Epub 2025 Apr 14. PMID 40227959
- [Background] Cai YH, Zhong JW, Ma HY, Szmuk P, Wang CY, Wang Z, Zhang XL, Dong LQ, Liu HC. Effect of Remimazolam on Emergence Delirium in Children Undergoing Laparoscopic Surgery: A Double-blinded Randomized Trial. Anesthesiology. 2024 Sep 1;141(3):500-510. doi: 10.1097/ALN.0000000000005077. PMID 38758221
- [Background] Badran BW, Brown JC, Dowdle LT, Mithoefer OJ, LaBate NT, Coatsworth J, DeVries WH, Austelle CW, McTeague LM, Yu A, Bikson M, Jenkins DD, George MS. Tragus or cymba conchae? Investigating the anatomical foundation of transcutaneous auricular vagus nerve stimulation (taVNS). Brain Stimul. 2018 Jul-Aug;11(4):947-948. doi: 10.1016/j.brs.2018.06.003. Epub 2018 Jun 6. No abstract available. PMID 29895444
- [Background] May SM, Reyes A, Martir G, Reynolds J, Paredes LG, Karmali S, Stephens RCM, Brealey D, Ackland GL. Acquired loss of cardiac vagal activity is associated with myocardial injury in patients undergoing noncardiac surgery: prospective observational mechanistic cohort study. Br J Anaesth. 2019 Dec;123(6):758-767. doi: 10.1016/j.bja.2019.08.003. Epub 2019 Sep 3. PMID 31492527
- [Background] Abbott TEF, Pearse RM, Cuthbertson BH, Wijeysundera DN, Ackland GL; METS study investigators. Cardiac vagal dysfunction and myocardial injury after non-cardiac surgery: a planned secondary analysis of the measurement of Exercise Tolerance before surgery study. Br J Anaesth. 2019 Feb;122(2):188-197. doi: 10.1016/j.bja.2018.10.060. Epub 2018 Dec 17. PMID 30686304
- [Background] Wang X, Huang ZG, Gold A, Bouairi E, Evans C, Andresen MC, Mendelowitz D. Propofol modulates gamma-aminobutyric acid-mediated inhibitory neurotransmission to cardiac vagal neurons in the nucleus ambiguus. Anesthesiology. 2004 May;100(5):1198-205. doi: 10.1097/00000542-200405000-00023. PMID 15114218
- [Background] May SM, Chiang E, Reyes A, Martir G, Patel A, Karmali S, Patel S, West S, Del Arroyo AG, Gourine AV, Ackland GL. Neuromodulation of innate immunity by remote ischaemic conditioning in humans: Experimental cross-over study. Brain Behav Immun Health. 2021 Jul 15;16:100299. doi: 10.1016/j.bbih.2021.100299. eCollection 2021 Oct. PMID 34589791
- [Background] Ackland GL, Abbott TEF, Cain D, Edwards MR, Sultan P, Karmali SN, Fowler AJ, Whittle JR, MacDonald NJ, Reyes A, Paredes LG, Stephens RCM, Del Arroyo AG, Woldman S, Archbold RA, Wragg A, Kam E, Ahmad T, Khan AW, Niebrzegowska E, Pearse RM. Preoperative systemic inflammation and perioperative myocardial injury: prospective observational multicentre cohort study of patients undergoing non-cardiac surgery. Br J Anaesth. 2019 Feb;122(2):180-187. doi: 10.1016/j.bja.2018.09.002. Epub 2018 Oct 2. PMID 30686303
- [Background] Sullere S, Kunczt A, McGehee DS. A cholinergic circuit that relieves pain despite opioid tolerance. Neuron. 2023 Nov 1;111(21):3414-3434.e15. doi: 10.1016/j.neuron.2023.08.017. Epub 2023 Sep 20. PMID 37734381
- [Background] Fang J, Rong P, Hong Y, Fan Y, Liu J, Wang H, Zhang G, Chen X, Shi S, Wang L, Liu R, Hwang J, Li Z, Tao J, Wang Y, Zhu B, Kong J. Transcutaneous Vagus Nerve Stimulation Modulates Default Mode Network in Major Depressive Disorder. Biol Psychiatry. 2016 Feb 15;79(4):266-73. doi: 10.1016/j.biopsych.2015.03.025. Epub 2015 Apr 2. PMID 25963932
- [Background] Han B, Li X, Hao J. The cholinergic anti-inflammatory pathway: An innovative treatment strategy for neurological diseases. Neurosci Biobehav Rev. 2017 Jun;77:358-368. doi: 10.1016/j.neubiorev.2017.04.002. Epub 2017 Apr 6. PMID 28392244
- [Background] Qi M, Huang Y, Mai R, Yan Z, Xu B, Liu B, Zhang Y. Baseline functional connectivity of the basal forebrain-cortical circuit predict taVNS treatment response in primary insomnia: a randomized controlled trial and fMRI study. BMC Med. 2025 Jul 9;23(1):412. doi: 10.1186/s12916-025-04126-7. PMID 40629377
- [Background] Austelle CW, Cox SS, Connolly DJ, Baker Vogel B, Peng X, Wills K, Sutton F, Tucker KB, Ashley E, Manett A, Cortese B, Short EB, Badran BW. Accelerated Transcutaneous Auricular Vagus Nerve Stimulation for Inpatient Depression and Anxiety: The iWAVE Open Label Pilot Trial. Neuromodulation. 2025 Jun;28(4):672-681. doi: 10.1016/j.neurom.2025.02.003. Epub 2025 Mar 19. PMID 40117415
- [Background] Zhang J, Chen Q, Shen Q, Yan C, Jiang T, Li J, Sayer S, Ai Z, Yu X, Zeng Q, Chen G. Effectiveness of Transcutaneous Auricular Vagal Nerve Stimulation on Alleviating Postoperative Pain Following Thoracoscopic Lobectomy: A Participant- and Assessor-blinded, Randomized Controlled Trial. Clin J Pain. 2025 Oct 1;41(10):e1315. doi: 10.1097/AJP.0000000000001315. PMID 40775700
- [Background] Ilfeld BM, Finneran JJ 4th, Alexander B, Abramson WB, Sztain JF, Ball ST, Gonzales FB, Abdullah B, Cha BJ, Said ET. Percutaneous auricular neuromodulation (nerve stimulation) for the treatment of pain following total knee arthroplasty: a randomized, double-masked, sham-controlled pilot study. Reg Anesth Pain Med. 2025 Jan 7;50(1):26-35. doi: 10.1136/rapm-2023-105028. PMID 38388019
- [Background] Patel ABU, Bibawy PPWM, Althonayan JIM, Majeed Z, Gan WL, Abbott TEF, Ackland GL. Effect of transauricular nerve stimulation on perioperative pain: a single-blind, analyser-masked, randomised controlled trial. Br J Anaesth. 2023 Apr;130(4):468-476. doi: 10.1016/j.bja.2022.12.025. Epub 2023 Feb 22. PMID 36822987
- [Background] Patel ABU, Weber V, Gourine AV, Ackland GL. The potential for autonomic neuromodulation to reduce perioperative complications and pain: a systematic review and meta-analysis. Br J Anaesth. 2022 Jan;128(1):135-149. doi: 10.1016/j.bja.2021.08.037. Epub 2021 Nov 18. PMID 34801224
- [Background] Patel A, Schieble T, Davidson M, Tran MC, Schoenberg C, Delphin E, Bennett H. Distraction with a hand-held video game reduces pediatric preoperative anxiety. Paediatr Anaesth. 2006 Oct;16(10):1019-27. doi: 10.1111/j.1460-9592.2006.01914.x. PMID 16972829
- [Background] Lee J, Lee J, Lim H, Son JS, Lee JR, Kim DC, Ko S. Cartoon distraction alleviates anxiety in children during induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1168-73. doi: 10.1213/ANE.0b013e31824fb469. Epub 2012 Sep 25. PMID 23011563
- [Background] Salonen M, Kanto J, Iisalo E, Himberg JJ. Midazolam as an induction agent in children: a pharmacokinetic and clinical study. Anesth Analg. 1987 Jul;66(7):625-8. PMID 3605671
- [Background] Kim YH, Yoon SZ, Lim HJ, Yoon SM. Prophylactic use of midazolam or propofol at the end of surgery may reduce the incidence of emergence agitation after sevoflurane anaesthesia. Anaesth Intensive Care. 2011 Sep;39(5):904-8. doi: 10.1177/0310057X1103900516. PMID 21970137
- [Background] Kawai M, Kurata S, Sanuki T, Mishima G, Kiriishi K, Watanabe T, Ozaki-Honda Y, Yoshida M, Okayasu I, Ayuse T, Tanoue N, Ayuse T. The effect of midazolam administration for the prevention of emergence agitation in pediatric patients with extreme fear and non-cooperation undergoing dental treatment under sevoflurane anesthesia, a double-blind, randomized study. Drug Des Devel Ther. 2019 May 17;13:1729-1737. doi: 10.2147/DDDT.S198123. eCollection 2019. PMID 31190751
- [Background] Cho EJ, Yoon SZ, Cho JE, Lee HW. Comparison of the effects of 0.03 and 0.05 mg/kg midazolam with placebo on prevention of emergence agitation in children having strabismus surgery. Anesthesiology. 2014 Jun;120(6):1354-61. doi: 10.1097/ALN.0000000000000181. PMID 24566243
- [Background] Hauber JA, Davis PJ, Bendel LP, Martyn SV, McCarthy DL, Evans MC, Cladis FP, Cunningham S, Lang RS, Campbell NF, Tuchman JB, Young MC. Dexmedetomidine as a Rapid Bolus for Treatment and Prophylactic Prevention of Emergence Agitation in Anesthetized Children. Anesth Analg. 2015 Nov;121(5):1308-15. doi: 10.1213/ANE.0000000000000931. PMID 26332857
- [Background] Lin Y, Chen Y, Huang J, Chen H, Shen W, Guo W, Chen Q, Ling H, Gan X. Efficacy of premedication with intranasal dexmedetomidine on inhalational induction and postoperative emergence agitation in pediatric undergoing cataract surgery with sevoflurane. J Clin Anesth. 2016 Sep;33:289-95. doi: 10.1016/j.jclinane.2016.04.027. Epub 2016 May 18. PMID 27555179
- [Background] Kim MS, Moon BE, Kim H, Lee JR. Comparison of propofol and fentanyl administered at the end of anaesthesia for prevention of emergence agitation after sevoflurane anaesthesia in children. Br J Anaesth. 2013 Feb;110(2):274-80. doi: 10.1093/bja/aes382. Epub 2012 Oct 26. PMID 23103775
- [Background] Gao Z, Zhang J, Nie X, Cui X. Effectiveness of Intravenous Ibuprofen on Emergence Agitation in Children Undergoing Tonsillectomy with Propofol and Remifentanil Anesthesia: A Randomized Controlled Trial. J Pain Res. 2022 May 12;15:1401-1410. doi: 10.2147/JPR.S363110. eCollection 2022. PMID 35592817
- [Background] Tan Y, Shi Y, Ding H, Kong X, Zhou H, Tian J. mu-Opioid agonists for preventing emergence agitation under sevoflurane anesthesia in children: a meta-analysis of randomized controlled trials. Paediatr Anaesth. 2016 Feb;26(2):139-50. doi: 10.1111/pan.12815. Epub 2015 Nov 28. PMID 26614352
- [Background] Carbo A, Tresandi D, Tril C, Fernandez-Rodriguez D, Carrero E. Usefulness of a virtual reality educational program for reducing preoperative anxiety in children: A randomised, single-centre clinical trial. Eur J Anaesthesiol. 2024 Sep 1;41(9):657-667. doi: 10.1097/EJA.0000000000002032. Epub 2024 Jun 24. PMID 38916221
- [Background] Byun S, Song S, Kim JH, Ryu T, Jeong MY, Kim E. Mother's recorded voice on emergence can decrease postoperative emergence delirium from general anaesthesia in paediatric patients: a prospective randomised controlled trial. Br J Anaesth. 2018 Aug;121(2):483-489. doi: 10.1016/j.bja.2018.01.042. Epub 2018 Apr 17. PMID 30032889
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Mason KP. Paediatric emergence delirium: a comprehensive review and interpretation of the literature. Br J Anaesth. 2017 Mar 1;118(3):335-343. doi: 10.1093/bja/aew477. PMID 28203739
- [Background] Abbas MS, El-Hakeem EEA, Kamel HE. Three minutes propofol after sevoflurane anesthesia to prevent emergence agitation following inguinal hernia repair in children: a randomized controlled trial. Korean J Anesthesiol. 2019 Jun;72(3):253-259. doi: 10.4097/kja.d.18.00345. Epub 2019 Mar 6. PMID 30841030
- [Background] He J, Zhang L, Tao T, Wen X, Chen D, Zheng X, Luo C, Liang H, Wang H. Nalbuphine reduces the incidence of emergence agitation in children undergoing Adenotonsillectomy: A prospective, randomized, double-blind, multicenter study. J Clin Anesth. 2023 May;85:111044. doi: 10.1016/j.jclinane.2022.111044. Epub 2022 Dec 23. PMID 36566649
- [Background] Yang X, Lin C, Chen S, Huang Y, Cheng Q, Yao Y. Remimazolam for the Prevention of Emergence Delirium in Children Following Tonsillectomy and Adenoidectomy Under Sevoflurane Anesthesia: A Randomized Controlled Study. Drug Des Devel Ther. 2022 Sep 30;16:3413-3420. doi: 10.2147/DDDT.S381611. eCollection 2022. PMID 36203819
- [Background] Wang Z, Wang X, Yang Y, He X, Jia W, Yao X, Sheng X, Jiao H. The effect of repeated maternal voice orientation on postoperative emergence agitation in children following tonsillectomy and adenoidectomy: A randomized controlled trial. J Clin Anesth. 2025 Jun;104:111851. doi: 10.1016/j.jclinane.2025.111851. Epub 2025 May 2. PMID 40318514
- See also: The First Affiliated Hospital of Zhejiang Chinese Medical University official site — https://www.zjhtcm1931.cn/

DOCUMENTS (3):
  • Study Protocol (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT07394647/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT07394647/SAP_001.pdf
  • Informed Consent Form (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT07394647/ICF_002.pdf